CLINICAL TRIAL: NCT02396654
Title: Accuracy of Five Dimensional Ultrasound Long Bones Fetal Biometry (5DUS LB ) for Prediction of Fetal Weight Compared to Two Dimensional Ultrasound: a Pilot Study
Brief Title: 5D LB Ultrasound in Determination of Fetal Weight in Normal Pregnancy : A Pilot Study
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dr mohamed laban, professor, Ain Shams University
Other Study IDs: m2492
Record Dates: First submitted 2015-03-19; First posted 2015-03-24 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Fetal Weight
MeSH Terms: conditions — Fetal Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- normal pregnant women: Normal pregnant women between 37 and 42 weeks gestation.
  Interventions: Other: 2D and 5D LB ultrasound comparison for fetal weight estimation

INTERVENTIONS:
Other: 2D and 5D LB ultrasound comparison for fetal weight estimation — 2D and 5DUS LB will be done for term pregnant women and fetal weight will be estimated by the hadlock formula. Accuracy of estimated fetal weight by both techniques will be compared to actual birth weight.

SUMMARY:
5D and 2D ultrasound will be done to normal pregnant women between 37 to 42 weeks gestation and fetal weight will be estimated using the hadlock formula using biometry measured by both ultrasounds. Accuracy of 5D ultrasound in determining fetal weight will be determined.

ELIGIBILITY:
Inclusion Criteria:

* 20-40years
* singleton pregnancy
* normal pregnancy

Exclusion Criteria:

* Intrauterine fetal death
* multiple pregnancy
* congenital anomaly
* nonvisualized fetal parts by ultrasound
* maternal medical disorders like diabetes and hypertension

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal pregnant women
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of 5D LB ultrasound in determining fetal weight (estimated by hadlock formula - Accuracy of estimated fetal weight by ultrasound will be compared to actual birth weight) | 48hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt